CLINICAL TRIAL: NCT01614340
Title: Treating Pain to Reduce Disability Among Older Home Health Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visiting Nurse Service of New York (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Weill Medical College of Cornell University (Other); Ithaca College (Other); Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HS020648-01A1 (AHRQ)
Record Dates: First submitted 2012-05-22; First posted 2012-06-07 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Arthritis - Post Surgical; Other Activity-limiting Pain
Keywords: Home care; Cognitive-Behavioral techniques; Physical Therapy; Pain; Older Adults
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other): Usual Physical Therapy Plan of Care
  Interventions: Behavioral: Cognitive-Behavioral Pain Self-management Program
- Usual Care Plus Pain Management Program (Other): Behavioral: Cognitive-Behavioral Pain Self-management Program.
  Interventions: Behavioral: Cognitive-Behavioral Pain Self-management Program

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Pain Self-management Program — The main study intervention is training of the PTs on teams randomized into the intervention group in the evidence-based CBPSM program which has been translated for use in home health care with patients who have activity-limiting pain. The program is designed to be implemented in a manner that allows for maximal integration into routine PT care of home health patients. This will be possible because the CBPSM techniques, together with exercise and other PT techniques that constitute customary PT care, are reciprocally reinforcing. Both treatments (CBPSM and PT) encourage the use of similar behavioral and pain self-management coping skills to enhance behavioral activation, perceptions of self-efficacy, self-control, and personal mastery with regard to the management of pain.

SUMMARY:
The overall goal of this real-world comparative effectiveness research (CER) study is to reduce disability among older home health patients by treating their pain more effectively. To achieve this goal the investigators will conduct a cluster randomized controlled trial of a physical therapist (PT) delivered intervention provided to VNSNY home health care patients with activity-limiting pain. The intervention is an evidence-based non-pharmacological program to reduce pain and pain-related disability that utilizes cognitive-behavioral pain self-management (CBPSM) techniques.

DETAILED DESCRIPTION:
This project will compare the effectiveness of usual care provided to older home health patients admitted with activity-limiting pain to usual care plus instruction by PTs in CBPSM techniques. The project also will examine differences in the effectiveness of the intervention among different race/ethnicity groups and individuals with different pain types, as well as the fidelity of intervention-group PTs to the CBPSM program.

The specific aims of this CER study that will include sizeable numbers of Hispanics, non-Hispanic African Americans and non-Hispanic white patients ages 55 and older are: (1) to compare the effectiveness of usual care provided to older home health patients admitted with activity-limiting pain to usual care plus instruction by PTs in CBPSM techniques; and (2) to examine the heterogeneity of CBPSM treatment effects among patients with different pain conditions and minority group status.

ELIGIBILITY:
Inclusion Criteria:

* VNSNY patient in the adult home healthcare program
* Services are being provided in the Bronx, Brooklyn, Manhattan, Queens, Staten Island, Nassau or Westchester
* VNSNY Plan of Care includes physical therapy
* Age 55 or older
* Speaks English
* Has a telephone
* Activity-limiting pain

Exclusion Criteria:

* Significant cognitive impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement on Performance-Based Measures of Functioning Among Intervention Patients | Baseline/Intake and 60 day follow up
  Patients receiving usual care plus the intervention when compared with participants receiving usual care only will demonstrate (1) Significantly better results as measured by the Timed Up and Go test; Timed Chair Stands, and Timed Foot Taps test;(2) Significantly better ADL functioning;(3) Significantly reduced levels of pain-related disability as measured by the Roland Morris Disability Questionnaire; and (4) Significantly reduced levels of pain intensity and increased levels of pain relief as measured by the Brief Pain Inventory.

SECONDARY OUTCOMES:
Lower Rates of Service Utilization Within Intervention Group | 60 day follow up survey
  Patients receiving the intervention plus usual care when compared to patients receiving usual care only will demonstrate significantly lower emergency department and hospital use during the follow-up period (as reported by the patient).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Murtaugh, PhD, Principal Investigator — Visiting Nurse Service of New York; Cary Reid, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Visiting Nurse Service of New York, New York, New York, United States

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5555786